CLINICAL TRIAL: NCT06440642
Title: The Effect of the Steep Trendelenburg Position on Intraocular Pressure ın Patients Undergoing Total Laparoscopic Hysterectomy
Brief Title: The Effect of the Steep Trendelenburg Position on Intraocular Pressure
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İrem DURMUS, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2023/51,1/250/33
Record Dates: First submitted 2024-05-23; First posted 2024-06-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Laparoscopic Surgery; Intraocular Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- steep trendelenburg: Patients Undergoing Laparoscopic Hysterectomy
  Interventions: Device: tonopen

INTERVENTIONS:
Device: tonopen — Intraoculer pressure will be measured in the supine position after intubation (T1), during pneumoperitoneum (T2), when placed in steep trendelenburg posıtıon (T3), at the end of the operation when pneumoperitoneum is terminated (T4), after being placed back in the supine position (T5), and 10 minutes after being placed back in the supine position (T6).

SUMMARY:
A total of 50 patients aged between 18-60 years, classified as American Society of Anesthesiologists (ASA) I-II, undergoing elective total laparoscopic hysterectomy in the steep trendelenburg position (STP) will be included in the study. Preoperatively, an ophthalmologist will perform an eye examination on the patients, and intraocular pressure will be measured using a non-contact computerized tonometer (Topcon CT-800, Japan). Central corneal thickness and iridocorneal angle will be measured using a topography device (Sirius Topography, CSO, Italy), and the thickness of the retinal nerve fiber layer (RNFL) will be measured using an optical coherence tomography (OCT) device (DRI OCT Triton, Topcon, Japan). Patients' demographic data and operation durations will be recorded. Intraocular pressure (IOP) will be measured in the supine position after intubation (T1), during pneumoperitoneum (T2), in the steep Trendelenburg position (23°, head down) (T3), at the end of the operation when pneumoperitoneum is terminated (T4), after returning to the supine position (T5), and 10 minutes after returning to the supine position (T6). Simultaneously with IOP measurements, the patients' hemodynamic data (Blood pressure, heart rate, end-tidal CO2, partial saturation) will be recorded.

DETAILED DESCRIPTION:
This study is planned to be conducted in the operating room of Kartal Dr. Lütfi Kırdar City Hospital between June 2024 and July 2024. A total of 50 patients aged between 18-60 years, classified as ASA I-II, undergoing elective total laparoscopic hysterectomy in the steep Trendelenburg position will be included in the study. Patients who are under 18 years or over 60 years, classified as ASA III or above, or have pre-existing eye conditions causing intraocular pressure changes such as glaucoma or ocular hypertension, cranial tumors, or any conditions that may be affected by increased intracranial pressure will not be included in the study.

All patients will undergo a preoperative evaluation the day before surgery, and written informed consent will be obtained for participation in the study. Patients who agree to participate will have an eye examination performed by an ophthalmologist preoperatively. Intraocular pressure (IOP) will be measured using a non-contact computerized tonometer (Topcon CT-800, Japan). Central corneal thickness and iridocorneal angle will be measured using a topography device (Sirius Topography, CSO, Italy), and the thickness of the retinal nerve fiber layer (RNFL) will be measured using an optical coherence tomography (OCT) device (DRI OCT Triton, Topcon, Japan).

Sure, here is the translation of your text into English:

---

The anesthesia protocol will be standardized for the drugs used during the procedure. Standard anesthesia induction will be provided with 2 mg IV midazolam, 3 mg/kg IV propofol, 100 mcg IV fentanyl, and 0.8 mg/kg IV rocuronium. Sevoflurane at 1 Minimum Alveolar Concentration (MAC) will be used for anesthesia maintenance. While the patient is in the supine position, intraperitoneal CO2 insufflation will be used to create pneumoperitoneum. The patients will then be placed in the steep Trendelenburg position (25 degrees from horizontal) at the maximum Trendelenburg angle (STP). All procedures will be performed in the same operating room, on the same table, and at the same angle. Intraperitoneal pressure will be maintained at 15 mm Hg throughout the surgery. At the end of the operation, patients will be awakened and transferred to the recovery unit. In the recovery unit, patients will be monitored for at least 30 minutes.

Intraocular pressure (IOP) will be measured in the supine position using a contact handheld tonometer (TONO-PEN AVIA, Reichert, USA). The Tono-pen is chosen for its speed, the ability to measure across multiple patients with single-use latex tip covers, ease of use, accuracy, and reliability in various positions. Five consecutive measurements will be taken for each eye. If the variability between consecutive measurements exceeds 5%, the measurements will be repeated. The average of the five measurements will be taken for each measurement. All measurements will be performed by the same ophthalmologist. All surgical operations will be conducted in the morning or early afternoon to prevent diurnal variations in IOP. All surgeries will be performed by the same surgical team.

The demographic data of the patients and the durations of the operations will be recorded. IOP will be measured in the supine position after intubation (T1), during pneumoperitoneum (T2), when placed in STP (23° head down) (T3), at the end of the operation when pneumoperitoneum is terminated (T4), after being placed back in the supine position (T5), and 10 minutes after being placed back in the supine position (T6). Simultaneously with IOP measurements, the patients' hemodynamic data (blood pressure, heart rate, end-tidal CO2, partial saturation) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* electively laparoscopic hysterectomy surgery with steep trendelenburg position
* ASA I-II
* Between 18-60 years old

Exclusion Criteria:

* Those under 18 or over 60 years old,
* ASA III and above,
* pre-existing eye conditions such as glaucoma, ocular hypertension, or other conditions affecting intraocular pressure
* those with conditions such as cranial tumors

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include 50 patients aged between 18 and 60 years with ASA I-II who will undergo elective total laparoscopic hysterectomy in the steep trendelenburg position.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluate patients' intraoculer pressure | during surgery and 10 minutes after the end of the operation
  the primary aim of the study is to evaluate patients' intraoculer pressure change during laparoscopic hysterectomy, position of steep trendelenburg

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lütfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided